CLINICAL TRIAL: NCT01935765
Title: Sleep Apnea in Type 1 Diabetes : Prevalence, Role of Glycemic Control and Autonomic Neuropathy
Brief Title: Sleep Apnea in Type 1 Diabetes
Acronym: DIASOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P111009
Record Dates: First submitted 2013-09-02; First posted 2013-09-05 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Type 1 Diabetes, Sleep Apnea Syndrome
Keywords: Type 1 diabetes, sleep apnea, polysomnography,; autonomic neuropathy, intima media thickness
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Sleep Apnea Syndromes | interventions — Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diabetes people (Experimental): 99 Type 1 diabetic patients aged 18 to 60 years, diagnosed since at least a year
  Interventions: Other: Polysomnography; Other: Evaluation of the autonomous nervous system; Other: Clinical examination of the sleep; Other: Clinical examination of diabetology; Other: Biological dosages; Other: Electrocardiogram (ECG); Other: Carotid echography; Other: Blood pressure
- healthy volunteers (controll group) (Experimental): 46 healthy volunteers matched by age, gender and body mass index
  Interventions: Other: Polysomnography; Other: Evaluation of the autonomous nervous system; Other: Clinical examination of the sleep; Other: Biological dosages; Other: Electrocardiogram (ECG); Other: Carotid echography; Other: Blood pressure

INTERVENTIONS:
Other: Polysomnography — Diabetes people: Examination diagnosis of the sleep apnea A night at the hospital
Other: Evaluation of the autonomous nervous system — blood pressure, Heart frequence, deep breath, Orthostatism, Vasalva, Low blood pressure orthostatic
Other: Clinical examination of the sleep — Functional signs, collection of medical histories and associated pathologies, Pittsburgh Sleep Quality Index PSQI, Functional Outcomes of Sleep Questionnaire FOSQ, Epworth Sleepiness Scale ESS, Hospital Anxiety and Depression scale HAD
Other: Clinical examination of diabetology — history of diabet, observance, ophthalmological, renal, macroangiopathic and neuronal complications, Toronto scale, Diabetes Quality of Life (DQOL) Questionnaire
  Arms: Diabetes people
Other: Biological dosages — Hematology, glycemia, lipids, CRP, creatinine, ferritin, glycosylated hemoglobin, transaminase, microalbuminuria, urine test
Other: Electrocardiogram (ECG) — Electrocardiogram (ECG)
Other: Carotid echography — Carotid echography
Other: Blood pressure — Blood pressure

SUMMARY:
Sleep apnea syndrome is strongly associated to type 2 diabet, partly and this is partly due to obesity. Treatment of sleep apnea may improve hypertension, cardiovascular risk and in some studies diabetes status. Few data are available for type 1 diabetes but suggest that the prevalence of sleep apnea syndrome may be high. We plan to compare the prevalence of sleep apnea syndrome assessed by polysomnography in a sample of type 1 diabetic patients and a control group matched by age, gender and body mass index. The secondary objective is to determine if the presence of an autonomic neuropathy or poorly controlled diabetes (assessed by glycosylated haemoglobin) may or not contribute to the presence of sleep apnea in the diabetic group.

DETAILED DESCRIPTION:
Diagnostic protocol designed to evaluate if if sleep apnea syndrome is more frequent in type 1 diabetes than in general population and therefore deserves to be more systematically suspected and actively diagnosed in this patients. Sleep apnea syndrome is a heavy burden as a matter of quality of life: it is responsible for fatigue, diurnal sleepiness, cognitive impairment, poor and /or non restorative sleep, morning headaches, depressive mood…Adequate treatment provides a rapid and, most of the time, complete relief of these symptoms.

On an other hand, Sleep Apnea is and independent risk factor for cardiovascular mortality and morbidity in young and middle aged subjects, also reversed by treatment. It might be therefore important for type 1 diabetic patients who have already an increased cardiovascular risk to be properly diagnosed for sleep apnea. A systematic screening for sleep apnea is already recommended for patients with type 2 diabetes by experts.

A secondary objective is to determine if the presence of a sleep apnea syndrome in type 1 diabetic patients is associated to an autonomic neuropathy, a poor glycemic control , a poorer quality of life , a poorer quality of sleep, more severe cardiovascular consequences and biological impairment.

ELIGIBILITY:
Inclusion Criteria:

* 99 Type 1 diabetic patients

  * man or woman aged 18 to 60 years
  * diagnosed since at least a year
  * having signed a consent
  * with in a national insurance scheme
* and 46 healthy volunteers matched by age , gender and body mass index

  * man or woman aged 18 to 60 years
  * having signed a consent
  * with in a national insurance scheme

Exclusion Criteria:

for both

* sleep apnea syndrome already known
* acute respiratory or cardiovascular disease
* impairment of consciousness
* sepsis
* cirrhosis
* hypnotic, opiate or psychotropic drug treatment 2 weeks ago
* Pregnant or breast-feeding woman
* Do not speak French
* Benefiting from a legal protective measure
* diabet 1 or 2 just for volunteers people

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Compare the prevalence of sleep apnea syndrome by polysomnography between type 1 diabetic patients and healthy volunteers | 3 months
  Determine if prevalence of the sleep apnea syndrome is more raised at the patient's diabetics of type 1 (DT1) than in the general population and to collect elements to specify the determiners of this association (presence of an autonomous neuropathy and glycemic balance).
  sleep apnea syndrome as defined by the International Classification of Sleep Disorders 2

SECONDARY OUTCOMES:
Precise if glycemic balance as defined by glycosylated hemoglobin<7% during the last three months is associated or not to sleep apnea syndrome | 3 months
  Compare diabetic subjects with or without sleep apnea regarding the rate of poorly controlled diabetes (determined by the level of glycosylated haemoglobin)
Precise if the presence of an autonomic neuropathy (positive at 2 tests) is associated or not to sleep apnea syndrome | 3 months
  Compare diabetic subjects with or without sleep apnea regarding presence of autonomic neuropathy determined by clinical assessment
Compare the patients with or without sleep apnea regarding consequences especially cardiovascular markers and coagulation factors | 3 months
  Compare diabetic subjects with or without sleep apnea regarding other cardiovascular risk factors and consequences (intima media thickness)
Determine if the presence of sleep apnea syndrome has an impact upon quality of life and diabetes complications, micro or macroangiopathy | 3 months
  Compare diabetic subjects with or without sleep apnea regarding quality of sleep
Precise clinical symptoms in DT1 patients with Sleep apnea syndrome | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Viot-Blanc, MD, Study Director — Lariboisiere Hospital, APHP; Pierre-Jean Guillausseau, MD, PhD, Principal Investigator — Lariboisiere Hopistal, APHP
Locations (1):
- Véronique Viot-Blanc, Paris, Île-de-France Region, France